CLINICAL TRIAL: NCT00769275
Title: Detection of Ischemia in Asymptomatic Diabetics
Acronym: DIAD
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Astellas Pharma US, Inc. (Industry)
Responsible Party: Frans J Th Wackers, MD, PhD, Yale University School of Medicine
Other Study IDs: DIAD; HIC #11312
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2008-10-09 (Estimated); Status verified 2008-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: silent ischemia; type 2 diabetes mellitus; screening; cardiac outcome; Prevalence silent myocardial ischemia; Cardiac outcome in screened and not-screened subjects
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Screening at start study with Adenosine vasodilator stress Tc-99m Sestamibi SPECT imaging
- 2: No screening

SUMMARY:
Asymptomatic subjects with Type 2 Diabetes Mellitus were randomized to either screening with Tc-99m sestamibi adenosine SPECT imaging or no screening. All patients will be followed for 5 years for the occurrence of cardiac death or non-fatal myocardial infarction.

The aims are:

1. To prospectively assess the prevalence of silent myocardial ischemia in asymptomatic subjects with Type 2 Diabetes Mellitus.
2. To identify on the basis of clinical and/or biochemical variables in a high-risk cohort in which screening for coronary artery disease is appropriate.
3. To assess progression of (silent) myocardial ischemia after 3 years.
4. To assess the occurence of cardiac death or nonfatal myocardial infarction during 5 years follow-up in screened and not screened subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years
* Type 2 diabetes mellitus

Exclusion Criteria:

* Angina or anginal equivalent
* Abnormal rest ECG (Q or ST depression)
* Known CAD
* Stress testing within the last 3 years

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asymptomatic patients with type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 1123 (Actual)
Dates: Start 2000-08; Primary Completion 2007-09 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of silent myocardial ischemia in subjects randomized to screening was 22%. | At study entry
At repeat stress imaging three years after recruitment 79% of subjects showed resolution of ischemia, whereas only 10% developed new ischemia. | 3 years after start
Overall cardiac event rate (cardiac death, myocardial infarction) was 3.0%, not different in screened and not screened cohort | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Frans J Wackers, MD, Study Chair — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Background] Wackers FJ, Young LH, Inzucchi SE, Chyun DA, Davey JA, Barrett EJ, Taillefer R, Wittlin SD, Heller GV, Filipchuk N, Engel S, Ratner RE, Iskandrian AE; Detection of Ischemia in Asymptomatic Diabetics Investigators. Detection of silent myocardial ischemia in asymptomatic diabetic subjects: the DIAD study. Diabetes Care. 2004 Aug;27(8):1954-61. doi: 10.2337/diacare.27.8.1954. PMID 15277423
- [Background] Wackers FJ, Chyun DA, Young LH, Heller GV, Iskandrian AE, Davey JA, Barrett EJ, Taillefer R, Wittlin SD, Filipchuk N, Ratner RE, Inzucchi SE; Detection of Ischemia in Asymptomatic Diabetics (DIAD) Investigators. Resolution of asymptomatic myocardial ischemia in patients with type 2 diabetes in the Detection of Ischemia in Asymptomatic Diabetics (DIAD) study. Diabetes Care. 2007 Nov;30(11):2892-8. doi: 10.2337/dc07-1250. Epub 2007 Aug 6. PMID 17682123
- [Derived] Young LH, Wackers FJ, Chyun DA, Davey JA, Barrett EJ, Taillefer R, Heller GV, Iskandrian AE, Wittlin SD, Filipchuk N, Ratner RE, Inzucchi SE; DIAD Investigators. Cardiac outcomes after screening for asymptomatic coronary artery disease in patients with type 2 diabetes: the DIAD study: a randomized controlled trial. JAMA. 2009 Apr 15;301(15):1547-55. doi: 10.1001/jama.2009.476. PMID 19366774